CLINICAL TRIAL: NCT00187421
Title: Graft Imaging to Improve Patency (GRIIP)
Brief Title: Using Intraoperative Coronary Bypass Graft Imaging to Improve Graft Patency
Acronym: GRIIP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Heart and Stroke Foundation of Ontario (Other)
Responsible Party: Principal Investigator, Stephen E. Fremes, Head , Division of Cardiac Surgery, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HSF NA 5530
Record Dates: First submitted 2005-09-14; First posted 2005-09-16 (Estimated); Last update posted 2012-12-12 (Estimated); Status verified 2012-12

CONDITIONS: Coronary Disease
Keywords: coronary disease; angiography; intraoperative care; vascular patency
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- 1 (No Intervention): Graft patency assessment by routine clinical assessment with/without intraluminal coronary probe
- 2 (Experimental): Graft patency assessment by indocyanine green angiography and transit-time flowmetry
  Interventions: Procedure: Indocyanine green intraoperative angiogram and transit-time flowmetry

INTERVENTIONS:
Procedure: Indocyanine green intraoperative angiogram and transit-time flowmetry — ICG graft angiography following each distal anastomosis, and imaging of proximal anastomoses after all grafts completed.
  transit time flowmetry performed on all grafts after all grafts completed.
  Other Names: Novadaq Spy System; Medtronic Medistem
  Arms: 2

SUMMARY:
The primary objective of the proposed study is to determine if a strategy of intraoperative patency assessment and graft revision can decrease the rate of graft occlusion or significant stenosis (>50%) at 6-12 weeks after coronary artery bypass grafting (CABG) versus traditional operative management without routine intraoperative patency assessment. Patency will be assessed with a new fluorescence angiography technique as well as ultrasonic transit-time flow measurement. We hypothesize that the strategy of intraoperative patency assessment and graft revision will significantly reduce the frequency of graft occlusion at 6-12 weeks in comparison to patients who do not have intraoperative patency assessment. We also hypothesize that the strategy of intraoperative patency assessment and graft revision will significantly reduce the frequency of 50-99% stenoses at 6-12 weeks in comparison to patients who do not have intraoperative patency assessment. We expect both groups will experience similar perioperative outcomes but hypothesize that patients receiving a strategy of intraoperative patency assessment and graft revision will experience improved long-term graft patency and freedom from late clinical events at 5-6 years post-operatively.

DETAILED DESCRIPTION:
The immediate and long term success of coronary surgery is dependent on the construction of a high quality anastomosis with a durable conduit to an appropriate target coronary vessel. Significant advances in medical therapy including early post-operative aspirin administration and increased use of arterial grafting have improved early, midterm and late graft patency. However, modern coronary bypass series continue to report perioperative graft occlusions rates as high as 11%. These very early graft failures have been predominantly ascribed to technical problems at graft anastomosis sites and may be preventable. New intraoperative graft assessment technologies have recently become available which can identify technical problems such that they can be repaired in the operating room. However, these techniques increase the length of the bypass operation and may have false positives, which may lead to unnecessary and potentially damaging graft revisions. The primary objective of the proposed study is to determine if a strategy of intraoperative patency assessment and graft revision can decrease the rate of graft occlusion or significant stenosis(>50%) at 6-12 weeks after coronary artery bypass grafting (CABG) versus traditional operative management without routine intraoperative patency assessment.

ELIGIBILITY:
Inclusion Criteria:

* isolated aortocoronary bypass surgery
* left ventricular ejection fraction >20%
* expect at least 2 bypass grafts

Exclusion Criteria:

* renal insufficiency (creatinine >180 umol/L)
* known allergy to indocyanine green contrast dye
* severe peripheral vascular disease precluding femoral access
* known allergy to radiographic contrast media
* women of childbearing potential
* co-morbid illness which precludes the use of follow-up angiography
* geographically inaccessible for follow-up angiography

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2005-07; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Graft occlusion determined by conventional angiography or CT angiography | 4 days to 4 months following surgery

SECONDARY OUTCOMES:
50-99% graft stenosis on postoperative graft angiography | 4 day to 4 months postoperatively
Mortality, myocardial infarction, low output syndrome | Perioperatively
Major cardiac adverse events | 1 year postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Stephen E Fremes, MD,MSc,FRCSC, Principal Investigator — Division of Cardiac and Vascular Surgery, Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

REFERENCES:
- [Result] Singh SK, Desai ND, Chikazawa G, Tsuneyoshi H, Vincent J, Zagorski BM, Pen V, Moussa F, Cohen GN, Christakis GT, Fremes SE. The Graft Imaging to Improve Patency (GRIIP) clinical trial results. J Thorac Cardiovasc Surg. 2010 Feb;139(2):294-301, 301.e1. doi: 10.1016/j.jtcvs.2009.09.048. Epub 2009 Dec 16. PMID 20006356